CLINICAL TRIAL: NCT01811602
Title: The Efficacy of Pelvic Floor Muscle Training in Gynecological Cancer Survivors: A Pilot Study
Brief Title: Gynecological Pelvic Floor Muscle Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H12-02473; F12-00262 (Other Grant/Funding Number: Physiotherapy Foundation of Canada)
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Urinary Incontinence
Keywords: Training; Physiotherapy; Pelvic floor muscles
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training (Other): Pelvic floor muscle training delivered by a physiotherapist with clinical expertise and training in treating pelvic floor dysfunction
  Interventions: Other: Training
- Usual Care Control (Other): Participants randomized to this arm will receive a 1-page educational pamphlet on pelvic floor muscle training, specifically Kegel exercises, which is equivalent to current standard care. Individuals randomized to this group will be placed on the clinic waiting list and be eligible for treatment following completion of the 12 week (end of study) measures.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Training — The participants randomized to the pelvic floor muscle training intervention will receive pelvic floor muscle training (0-12 weeks) delivered by a physiotherapist with clinical expertise and training in treating pelvic floor dysfunction. The intervention is 9 individual, one-on-one, 45-minute sessions; weekly for weeks 0-6 and bi-weekly for weeks 7-12 (first session will be 60 minutes). The sessions will provide pelvic floor muscle training based on the latest evidence, including biofeedback, to teach the correct technique for pelvic floor contractions, and participants will be asked to complete daily pelvic floor exercises at home.
  Other Names: Pelvic Floor Muscle Training
  Arms: Training
Other: Usual Care — The participants randomized to the educational pamphlet intervention (usual care control) will receive a 1-page sheet on pelvic floor muscle training, specifically Kegel exercises, which is equivalent to current standard care. Individuals randomized to this group will be placed on the clinic waiting list and be eligible for treatment following completion of the 12 week (end of study) measures.
  Other Names: Educational pamphlet
  Arms: Usual Care Control

SUMMARY:
A randomized controlled trial pilot study to test the efficacy of a pelvic muscular training intervention led by a physiotherapist on urinary incontinence, quality of life and sexual health in women who report urinary urgency and incontinence following surgery and radiation treatment for gynecological cancer vs. usual care (a 1-page sheet on Kegel exercises).

ELIGIBILITY:
Inclusion Criteria:

- treated with surgery and adjuvant treatment, including radiation, for gynecological cancer within the last 3 years

Exclusion Criteria:

* stage IV cancer or stage III and IV cervical cancer
* radiation not part of treatment
* known spinal or long bone metastases diagnosis with a neuromuscular disorder that may impact pelvic floor muscle function
* urinary incontinence issues prior to cancer diagnosis
* scheduled or previous surgical treatment of incontinence
* fecal incontinence
* body mass index (BMI) > 35
* use of medications to improve bladder function
* unable to complete questionnaires in English or unable to actively participate in physiotherapy treatment provided in English.

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence | 12 weeks
  Urinary incontinence, measured using the International Consultation on Incontinence Questionnaire Urinary Incontinence (ICIQ-UI Short Form) and bladder diary

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Campbell, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Women's Health Centre, Vancouver, British Columbia, Canada